CLINICAL TRIAL: NCT06137404
Title: A Comparison of Metacarpophalangeal Joint Blocking Splint With Relative Motion Extension Splint for Trigger Finger
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Waikato Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: WaikatoH
Record Dates: First submitted 2023-10-29; First posted 2023-11-18 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Trigger Finger
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Splints

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Splint M (Active Comparator): Metacarpophalangeal joint blocking splint
  Interventions: Other: Splint
- Splint R (Experimental): Relative motion extension splint
  Interventions: Other: Splint

INTERVENTIONS:
Other: Splint — Comparison of splints for trigger finger

SUMMARY:
The purpose of this research is to evaluate the effectiveness of two splint designs in conservative management of trigger finger.

DETAILED DESCRIPTION:
This study aims to analyse and compare the effectiveness of metacarpophalangeal joint blocking splint versus relative motion extension splint for trigger finger. This will help us find out which one of the two splint designs is more effective in the management of trigger finger, thus improving treatment outcomes for patients with trigger finger.

ELIGIBILITY:
Inclusion Criteria:

* Trigger finger patient

Exclusion Criteria:

* Diabetes, non-English speaking

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Green's classification for trigger finger | 12 weeks
  Green's classification is an objective outcome measure. The therapist grades the triggering by observing the finger when the patient makes a full fist.
  Grade I: Pain/history of catching Grade II: Demonstrable catching but can actively extend digit Grade III: Demonstrable locking, requiring passive extension Grade IV: Fixed flexion contracture
  Lowest score is I; highest score is IV

SECONDARY OUTCOMES:
QuickDASH (Disability of Arm, Shoulder and Hand) | 12 weeks
  The QuickDASH is a patient rated questionnaire that rates patient's ability to perform certain tasks as well as severity of symptoms. The best score is 0 (no difficulty) and the lowest score is 100 (severe difficulty).

OTHER OUTCOMES:
Visual Analogue Scale (VAS) | 12 weeks
  The VAS is a patient rated outcome measure that enables the patient to rate the intensity of pain from 0 (no pain) to 10 (worse pain that can possibly be)

CONTACTS AND LOCATIONS:
Overall Officials: Aarti Parekh, B.Physio, Principal Investigator — Waikato Hospital
Locations (1):
- Waikato Hospital, Hamilton, Waikato Region, New Zealand